CLINICAL TRIAL: NCT03381326
Title: Biomarkers Study: Circulating Tumor Cells (CTC), Free DNA, Stem Cells and Epithelial-mesenchymal-transition (EMT) Related Antigens as Biomarkers of Activity of Cabazitaxel in Castration-resistant Prostate Cancer (CRPC): a Proof of Concept.
Brief Title: CTC, Free DNA, Stem Cells and EMT-related Antigens as Biomarkers of Activity of Cabazitaxel in CRPC.
Acronym: IRSTB030
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IRSTB030
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer; Metastatic Cancer; Castration-resistant Prostate Cancer; Circulating Tumor Cells
Keywords: circulating tumor cells; Castration-resistant Prostate Cancer; cabazitaxel; biomarker; free DNA; stem cells; EMT related antigens
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples and FFPE samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: blood and FFPE sample collection — blood sample and Formalin-fixed paraffin-embedded (FFPE) sample collection

SUMMARY:
Identification of biomarkers (Circulating Tumor Cells (CTC), free DNA, Stem Cells and EMT-related antigens) that may be predictive of outcome of activity of cabazitaxel treatment in castration-resistant prostate cancer.

DETAILED DESCRIPTION:
Circulating Tumor Cells, free DNA, Stem Cells and EMT-related antigens as biomarkers of activity of cabazitaxel in castration-resistant prostate cancer

Primary objectives: To evaluate the prognostic role of response of the copy number of androgen receptor (AR) and Phosphatase and tensin homolog (PTEN) and AR-V7 and other gene expression biomarkers in CTC and the investigators will compare these results with those obtained in plasma cell free DNA and RNA.

Eligible patients must have histologically or cytologically confirmed prostate cancer or unequivocal increased PSA . Metastatic and/or inoperable disease and received prior therapy with docetaxel and candidate to cabazitaxel treatment.

All patients receive cabazitaxel at standard schedule 25 mg/m2 q21. Blood sample will be collected for CTC evaluation at baseline, after the first cycle of therapy (optional), at first radiological evaluation (after 3 months), at disease progression (optional) or after 9-12 months of treatment for patients who did not show disease progression (optional). Disease progression defined according to Prostate Cancer Working Group 2 (PCWG2) criteria. On blood samples from Castration-Resistant Prostate Cancer (CRPC) patients the investigators will investigate the presence of the previously presented CTC, DNA and RNA free markers.

As an option, it will be possible to require a sample of the tumor collected during prostate surgery or during the biopsy.

All patients will be treated and monitored according to the local clinical practice. No additional procedures/patient visits in comparison with the usual clinical practice are planned for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document
2. Male aged >18 years with metastatic castration-resistant disease with documented clinical (imaging) and/or biochemical progression (PSA increasing values) during or after a previous docetaxel-based chemotherapy
3. Patients must have metastatic and/or inoperable disease
4. Patients must have received prior therapy docetaxel based and must be candidate to cabazitaxel
5. Life expectancy of greater than 3 months
6. Eastern Cooperative Oncology Group (ECOG) performance status <2

Exclusion Criteria:

1. Participants who are unable to provide informed consent
2. Participation in another clinical trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with castration-resistant prostate cancer
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 36 months
  time between the start of cabazitaxel and the ﬁrst date of progression as measured by PCWG-2 criteria.

SECONDARY OUTCOMES:
Overall survival (OS) | 36 months
  The overall survival will be calculated from date of the start of cabazitaxel to death

CONTACTS AND LOCATIONS:
Overall Officials: Ugo De Giorgi, Principal Investigator — Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST)
Locations (9):
- Italy (9):
  - Ospedali Riuniti Umberto I, Ancona, AN
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC
  - IRCCS AOU San martino IST, Genova, GE
  - Ospedale Civile degli Infermi, Rimini, RN
  - Azienda Ospedaliera Cannizzaro, Catania
  - Ospedale Maggiore della Carità, Novara
  - Istituto Oncologico del Veneto (IOV) - Università di Padova, Padua
  - Policlinico Universitario Campus Bio-Medico, Roma
  - Ospedale Sacro Cuore Don Calabria (Negrar), Verona

REFERENCES:
- [Derived] Gurioli G, Conteduca V, Brighi N, Scarpi E, Basso U, Fornarini G, Mosca A, Nicodemo M, Banna GL, Lolli C, Schepisi G, Ravaglia G, Bondi I, Ulivi P, De Giorgi U. Circulating tumor cell gene expression and plasma AR gene copy number as biomarkers for castration-resistant prostate cancer patients treated with cabazitaxel. BMC Med. 2022 Jan 31;20(1):48. doi: 10.1186/s12916-022-02244-0. PMID 35101049
- [Derived] Conteduca V, Wetterskog D, Castro E, Scarpi E, Romero-Laorden N, Gurioli G, Jayaram A, Lolli C, Schepisi G, Wingate A, Casadei C, Lozano R, Brighi N, Aragon IM, Marin-Aguilera M, Gonzalez-Billalabeitia E, Mellado B, Olmos D, Attard G, De Giorgi U. Plasma androgen receptor and response to adapted and standard docetaxel regimen in castration-resistant prostate cancer: A multicenter biomarker study. Eur J Cancer. 2021 Jul;152:49-59. doi: 10.1016/j.ejca.2021.04.025. Epub 2021 May 30. PMID 34077818